CLINICAL TRIAL: NCT01067690
Title: Phase II Trial for the Treatment of Advanced Classical Kaposi's Sarcoma With the HIV Protease Inhibitor Indinavir in Combination With Chemotherapy
Brief Title: Treatment With Indinavir and Chemotherapy for Advanced Classical Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ensoli, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Barbara Ensoli, MD, PhD, MD, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CKS/IND-CX/05
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Kaposi's Sarcoma
Keywords: classical Kaposi's sarcoma; chemotherapy; indinavir; HIV protease inhibitor; Advanced classical (non HIV-associated) Kaposi's sarcoma
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — Indinavir; Association

INTERVENTIONS:
Drug: Indinavir in association with Vinblastina +/- Bleomicina — Treatment consists in an induction phase where daily Indinavir (800 mg x 2/die, orally) will be combined together with systemic Vinblastine (10 mg intravenously) +/- Bleomycin (15 mg intramuscularly) in cycles administered every 3 weeks. As maximal response will occur, patients will undergo 2 additional Vinblastine +/- Bleomycin (consolidation) cycles upon continuous treatment with Indinavir. This will be followed by a maintenance phase with Indinavir alone (800 mg x 3/die, orally) in responder patients.

SUMMARY:
The purpose of this study is to determine the clinical response to daily Indinavir oral administration in association with a conventional chemotherapy based on cycles of systemic Vinblastine +/- Bleomycin in patients affected by advanced classical (non HIV-associated) Kaposi's sarcoma

DETAILED DESCRIPTION:
It has been recently demonstrated that HIV protease inhibitors (HIV-PI) exert direct anti-angiogenic and anti-tumor actions by blocking endothelial and tumor cell invasion and matrix metalloprotease (MMP) activity. Based on this data, we have started a phase II trial for the treatment of HIV-negative patients with CKS with the HIV-PI Indinavir. Indinavir was well tolerated and induced KS regression/improvement in early-stage disease, and prolonged stabilization in late-stage KS. Response required high plasma drug concentrations indicating a "therapeutic" drug threshold, and was associated with a decrease of circulating endothelial cells (CEC), basic fibroblast growth factor and MMP2 plasma levels. However, large, confluent tumor masses were generally not responsive (Monini et al, AIDS 2009). Thus, advanced KS may benefit at best by treatment with IND upon tumor debulking by conventional chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of KS
* Negative HIV ELISA test
* Being classified as stage III or IV
* Age ≥18 years
* Having interrupted any other anti-KS therapy since at least 2 weeks
* Being informed about the nature of the study and having signed the informed consent

Exclusion Criteria:

* Inability to give informed consent
* Presence of other concomitant diseases, neoplasia (excluding cutaneous tumors with limited extension and without diagnosis of melanoma) or any other life-threatening clinical condition that would compromise its compliance to the protocol
* Concomitant treatments (within 2 weeks prior to the study) with systemic immunomodulatory agents (i.e. glucocorticoids used as immunosuppressive agents, interferons) or chemotherapy
* Pregnancy
* Monolateral nephropathy or history of nephrolithiasis during the last 5 years
* Any clinically relevant and persistent alteration of laboratory values observed during screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
to determine the rate of complete responses at the end of treatment (including the maintenance phase) and of clinical responses after the maintenance phase, considering the residual debulked tumour (after the induction phase) as the reference point.

SECONDARY OUTCOMES:
to determine time to tumor progression, treatment tolerability, indinavir pharmacokinetic profile, biological markers of response (ie. angiogenesis and immunoactivation parameters, HHV8 viral load and immune response)

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Brambilla, MD, Principal Investigator — Dermatologic Unit, Ospedale Maggiore Policlinico, Milan, Italy
Locations (1):
- Dermatologic Unit, Ospedale Maggiore Policlinico, Milan, Italy, Milan, Italy, Italy

REFERENCES:
- [Background] Ensoli B, Sturzl M, Monini P. Cytokine-mediated growth promotion of Kaposi's sarcoma and primary effusion lymphoma. Semin Cancer Biol. 2000 Oct;10(5):367-81. doi: 10.1006/scbi.2000.0329. PMID 11100885
- [Background] Sgadari C, Barillari G, Toschi E, Carlei D, Bacigalupo I, Baccarini S, Palladino C, Leone P, Bugarini R, Malavasi L, Cafaro A, Falchi M, Valdembri D, Rezza G, Bussolino F, Monini P, Ensoli B. HIV protease inhibitors are potent anti-angiogenic molecules and promote regression of Kaposi sarcoma. Nat Med. 2002 Mar;8(3):225-32. doi: 10.1038/nm0302-225. PMID 11875492
- [Background] Sgadari C, Monini P, Barillari G, Ensoli B. Use of HIV protease inhibitors to block Kaposi's sarcoma and tumour growth. Lancet Oncol. 2003 Sep;4(9):537-47. doi: 10.1016/s1470-2045(03)01192-6. PMID 12965274
- [Background] Monini P, Sgadari C, Toschi E, Barillari G, Ensoli B. Antitumour effects of antiretroviral therapy. Nat Rev Cancer. 2004 Nov;4(11):861-75. doi: 10.1038/nrc1479. PMID 15516959
- [Background] Monini P, Sgadari C, Grosso MG, Bellino S, Di Biagio A, Toschi E, Bacigalupo I, Sabbatucci M, Cencioni G, Salvi E, Leone P, Ensoli B. Clinical course of classic Kaposi's sarcoma in HIV-negative patients treated with the HIV protease inhibitor indinavir. AIDS. 2009 Feb 20;23(4):534-8. doi: 10.1097/QAD.0b013e3283262a8d. PMID 19169139